CLINICAL TRIAL: NCT04327141
Title: Comparison of Protein Pacing, Intermittent Fast vs. Heart Healthy Diet on Body Weight and Composition, Cardiometabolic, Mood, and Gut Microbiome Health, in Overweight Men and Women During Weight Loss; 24 Months Follow-up Case Study of 100 Pound Weight Loss in a Male Study Participant
Brief Title: Low Sugar Protein Pacing, Intermittent Fasting Diet in Men and Women
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Skidmore College (Other)
Collaborators: Arizona State University (Other); Isagenix International LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1911-859
Record Dates: First submitted 2020-03-06; First posted 2020-03-30 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Weight Loss; Gut Microbiome; Anti-Aging
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Intervention Model Description: 40 overweight/obese adult men (n=20) and women (n=20) will be quasi-randomized to one of the two groups matched by sex (men/women) and body weight. Participants will be enrolled in the study as a single cohort and participate in a 8-week weight loss (WL) trial consisting of a single dietary intervention phase. A single male participant from the original P-IF group will continue following the identical P-IF from the original 4-8 week phase and 12 month follow up period (5-6 days of P; 1-2 day of IF) for an additional 12 month period (beyond the initial 12 monthfollow up case study period). The participant will consume the identical P-IF meal plan as the original 8 week study and 24 month follow up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Protein pacing and intermittent fasting (Experimental): During the 8-week weight loss (WL) phase, participants assigned to the P-IF will consist of P days, whereby female participants will consume four and male participants will consume five meals/snacks total, two of which (breakfast and lunch) will include a protein powder meal replacement mixed with water (240-400 kcals per meal) along with an evening dinner meal (~500 kcals), an afternoon snack (men only), and an evening snack (250 kcals). Subjects will be calorie restricted to ~1500 and ~1800 calories per day, women and men, respectively during P days. For each IF day, subjects will be provided a variety of supplements/snacks made by Isagenix International LLC. The P-IF group will be further divided into two subgroups for weeks 1-4. One subgroup will consist of five days of P and two days of IF, and the second subgroup will consist of six days of P and one day of IF. For weeks 5-8 both subgroups will follow 6 days of a P diet and 1 day IF.
  Interventions: Behavioral: P-IF
- Heart Healthy (Experimental): The HH group will observe the dietary guidelines in compliance with the National Cholesterol Education Program Therapeutic Lifestyle Changes (TLC) diet. This diet consists of consuming <35% of kcal as fat; 50%-60% of kcal as carbohydrates; <200 mg/dL of dietary cholesterol; and 20-30 g/day of fiber. The total calorie intake will be 1200 and 1500 calories per day, women and men, respectively during the weight loss phase (weeks 0-8).
  Interventions: Behavioral: HH

INTERVENTIONS:
Behavioral: P-IF — Protein pacing and intermittent fasting
  Arms: Protein pacing and intermittent fasting
Behavioral: HH — Heart Healthy
  Arms: Heart Healthy

SUMMARY:
This study will systematically quantify the effects of protein pacing and intermittent fasting (P-IF) on total and regional (abdominal) body composition (lean mass and fat mass), blood glucose and lipids, and anti-aging biomarkers, hunger ratings, and the gut microbiome in 40 overweight/obese adult men (n=20) and women (n=20) following a 8-week weight loss intervention. Participants will be enrolled in the study as a single cohort and participate in a 8-week weight loss (WL) trial consisting of a single dietary intervention phase. The purpose of the additional 12 month follow up case study (in addition to the initial 12-month case study period) is to scientifically document a significant weight loss and improved body composition following combined protein pacing intermittent fasting nutrition and a safe, effective exercise program in a study participant who achieved successful weight loss maintenance during the previous 12 month follow up study period.

DETAILED DESCRIPTION:
Previous research has shown combined protein pacing and intermittent fasting (PP-IF; 1-2 days per week) combined with moderate (20-30%) caloric restriction (CR) favorably enhance weight loss, body composition, cardiometabolic disease risk, oxidative stress, and toxin levels compared to a heart healthy diet in obese individuals following both weight loss and weight loss maintenance (Arciero et al. 2016; He et al. 2017; Zuo et al. 2016). However, less is known about whether a low sugar intake with this dietary pattern induces other significant health improvements, such as enhanced brain health (mood state), as well as gut microbiome and anti-aging indices, compared to a heart healthy diet. The novelty of the current proposal is of particular relevance and importance given the heightened popularity of low sugar dietary patterns shown to enhance health status. Most notably, among these low sugar diets touting the health benefits, are the ketogenic, paleolithic and Mediterranean diets. In addition, there is a great deal of public health emphasis on reducing overall carbohydrate intake, especially simple sugars, to improve cardiometabolic, gut, and body composition health. The dangers of high simple sugar intake are numerous, including increased risk for cardiometabolic disease (high blood lipids, hyperglycemia, insulin resistance, systemic inflammation, oxidative stress, obesity, elevated visceral fat, etc.). Thus, improvements in body composition and reductions in disease risk provides compelling evidence to pursue this study with vigor so as to generate a viable and healthy weight and fat loss strategy over the long term. Another major factor to augment long-term (>1 year) weight loss success, is inclusion of a safe and realistic exercise program (4 days/week) consisting of walking, stretching, and simple body weight movements such as sit-ups and push-ups. To date, there are no documented case studies of a human participant achieving a one hundred pound plus weight loss using protein pacing and intermittent fasting combined with a proven, safe and time-efficient exercise program.

The purpose of this study is to compare the effects of a low sugar protein pacing, intermittent fasting (P-IF) diet versus a heart healthy (HH) diet on indices of body weight, total and regional body composition, mood state, anti-aging, and cardiometabolic outcomes, and the gut microbiome during weight loss (0-8 weeks). Specifically, this study aims to compare a P-IF diet comprised of a calorie-restricted (1500 calories/day women; 1800 calories/day men) protein pacing diet (P, 4 meals/day women, 5 meals/day men) followed by a fast (IF, ~350-450 kcals/day) compared to an established calorie-restricted (1200 calories/day for women; 1500 calories/day men) heart healthy (HH) diet. The P-IF group will be divided into two subgroups for weeks 1-4. One subgroup will consist of five days of P and two days of IF, and the second subgroup will consist of six days of P and one day of IF. For weeks 5-8 both subgroups will follow 6 days of a P diet and 1 day IF. The purpose of the additional 12 month follow up case study (in addition to the initial 12-month case study period) is to scientifically document a significant weight loss and improved body composition following combined protein pacing intermittent fasting nutrition and a safe, effective exercise program in a study participant who achieved successful weight loss maintenance during the previous 12 month follow up study period.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking, healthy, but overweight/obese men and women with no known cardiovascular or metabolic diseases as assessed by a medical history and a comprehensive medical examination by their physicians
* Sedentary or lightly active (<30 min, 2d/wk of structured physical activity) as assessed by a Physical Activity questionnaire
* Overweight or obese (BMI>27.5 kg/m2; % body fat>30%)
* Weight stable (+/-2kg) for at least 6 months prior to beginning the study

Exclusion Criteria:

* Type II Diabetes
* Emphysema
* Significant heart disease (CABG, CHF, VFib, Hypercholesterolemia, Uncontrolled High Blood Pressure, etc.)
* COPD
* Cancer or undergoing treatment for cancer
* Allergies to milk or milk products, sugar alcohols, fructose, or gluten
* Anorexia or Bulimia
* Fasting intolerances/hypoglycemia
* Pregnant or plan to become pregnant during 8-week study

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-09-03 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in body weight | 0 weeks, 4 weeks, 8 weeks and monthly intervals during the 2 year Case Study
  Total body weight measurement

SECONDARY OUTCOMES:
Change in total and regional body fat and lean body mass | 0 weeks, 8 weeks, 1 year and 2 year of the Case study
  Quantitative measure of total body fat and lean mass using iDXA (dual x-ray absorptiometry)
Changes in feelings of hunger, fullness, satiety scores measured with a visual analog scale | 0 weeks, 4 weeks, 8 weeks and monthly intervals during the 2 year Case Study
  Hunger ratings using a visual analog scale ranging from 0-100 mm. A score closer to 0mm indicates no level of hunger related feelings and a score of 100 mm indicates extreme hunger-related feelings
Change in blood lipid levels | 0 weeks, 4 weeks, 8 weeks and every 6 months during the 2 year Case Study
  Venipuncture blood draw of 5ml per visit (weeks 0 and 8) and a single finger stick* of 40ul (week 4); *Finger stick at week 4 will only measure glucose and blood lipids
Change in gut microbiome, gastrointestinal symptoms, stool | 0 weeks, 4 weeks, 8 weeks and two month intervals during the 2 year Case Study
  Fecal gut microbiome communities will be sequenced using microbial DNA extracted from samples at 0, 4, and 8 weeks for each study arm. Amplified copies of the 16S rRNA gene will be evaluated for treatment differences in alpha (within-sample richness and evenness) and beta diversity (between-sample community structure). Relative and differential abundance of individual microbial taxa will also be measured. In addition, GI symptoms will be assessed using the Gastrointestinal symptom questionnaire and stool quality will be assessed with the Bristol stool chart
Change in blood pressure | 0 weeks, 4 weeks, 8 weeks and monthly intervals during the 2 year Case Study
  Quantitative measure of blood pressure using automated blood pressure monitor called a mobiligraph for 1 minute
Change in heart rate | 0 weeks, 4 weeks, 8 weeks and monthly intervals during the 2 year Case Study
  Quantitative measure of heart rate using automated heart rate monitor called a mobiligraph for 1 minute
Change in fat mass and muscle mass | 0 weeks, 4 weeks, 8 weeks and monthly intervals during the 2 year Case Study
  Quantitative measure of total body fat and muscle mass using BODPod (air displacement plethysmography)
Change in physical activity | 0 weeks, 4 weeks, 8 weeks, and monthly intervals during the 2 year of the Case study
  Quantitative measure of physical activity (kilocalories per day) using the ActiGraph accelerometer
Change in energy intake | 0 weeks, 4 weeks, 8 weeks, and monthly intervals during the 2 year of the Case study
  Quantitative measure of energy intake (kilocalories per day) using the 2-day food diary

CONTACTS AND LOCATIONS:
Overall Officials: Paul J Arciero, PhD, Principal Investigator — Skidmore College
Locations (1):
- Human Nutrition and Metabolism Laboratory, Saratoga Springs, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arciero PJ, Edmonds R, He F, Ward E, Gumpricht E, Mohr A, Ormsbee MJ, Astrup A. Protein-Pacing Caloric-Restriction Enhances Body Composition Similarly in Obese Men and Women during Weight Loss and Sustains Efficacy during Long-Term Weight Maintenance. Nutrients. 2016 Jul 30;8(8):476. doi: 10.3390/nu8080476. PMID 27483317
- [Background] He F, Zuo L, Ward E, Arciero PJ. Serum Polychlorinated Biphenyls Increase and Oxidative Stress Decreases with a Protein-Pacing Caloric Restriction Diet in Obese Men and Women. Int J Environ Res Public Health. 2017 Jan 10;14(1):59. doi: 10.3390/ijerph14010059. PMID 28075418
- [Background] Zuo L, He F, Tinsley GM, Pannell BK, Ward E, Arciero PJ. Comparison of High-Protein, Intermittent Fasting Low-Calorie Diet and Heart Healthy Diet for Vascular Health of the Obese. Front Physiol. 2016 Aug 29;7:350. doi: 10.3389/fphys.2016.00350. eCollection 2016. PMID 27621707
- [Derived] Mohr AE, Sweazea KL, Bowes DA, Jasbi P, Whisner CM, Sears DD, Krajmalnik-Brown R, Jin Y, Gu H, Klein-Seetharaman J, Arciero KM, Gumpricht E, Arciero PJ. Gut microbiome remodeling and metabolomic profile improves in response to protein pacing with intermittent fasting versus continuous caloric restriction. Nat Commun. 2024 May 28;15(1):4155. doi: 10.1038/s41467-024-48355-5. PMID 38806467
- [Derived] Mohr AE, Jasbi P, Bowes DA, Dirks B, Whisner CM, Arciero KM, Poe M, Gu H, Gumpricht E, Sweazea KL, Arciero PJ. Exploratory analysis of one versus two-day intermittent fasting protocols on the gut microbiome and plasma metabolome in adults with overweight/obesity. Front Nutr. 2022 Oct 26;9:1036080. doi: 10.3389/fnut.2022.1036080. eCollection 2022. PMID 36386914
- [Derived] Arciero PJ, Arciero KM, Poe M, Mohr AE, Ives SJ, Arciero A, Boyce M, Zhang J, Haas M, Valdez E, Corbet D, Judd K, Smith A, Furlong O, Wahler M, Gumpricht E. Intermittent fasting two days versus one day per week, matched for total energy intake and expenditure, increases weight loss in overweight/obese men and women. Nutr J. 2022 Jun 4;21(1):36. doi: 10.1186/s12937-022-00790-0. PMID 35658959